CLINICAL TRIAL: NCT03986957
Title: Novel Approaches of Advanced Neuroimaging Based on MRI Fiber Tracking to Detect Early Signs of Vascular Cognitive Impairment in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Collaborators: IRCCS Multimedica (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, Full Professor, MD, PhD, Neuromed IRCCS
Other Study IDs: LMB07
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Hypertension
Keywords: Vascular Cognitive Impairment; Magnetic Resonance Imaging; Blood Pressure Variability
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine for biochemical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensive patients: Patients with SBP: 140-159; DBP: 90-99
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions - observational study

SUMMARY:
Hypertension is the major risk factor for vascular cognitive impairment (VCI). One of the main limitations in the clinical approach to VCI is that, by the time that it is manifested, it might be too late to reverse the neurodegenerative process. Thus, early identification of predictive signs of later dementia is demanding for management of hypertensive patients (HT).This aim claims for new methods that compute in a cloud all possible data sources coming from patients (brain imaging, cognitive profile, clinical data), to extract discriminative aggregate biomarkers. Thus, this study aims at: 1) characterizing the predictive potential of an aggregate biomarker for dementia in HT, based on brain imaging, clinical and cognitive assessment; 2) evaluating the impact of blood pressure variability, besides systolic/diastolic blood pressure, on the progression of the aggregate biomarker; 3) assessing whether specific classes of antihypertensive drugs differently affect the progression of the aggregate biomarker. In order to do this, this study proposes to evaluate advanced brain imaging and cognitive profile in a cohort of hypertensive patients, at baseline and after a 1 year follow up, to identify an innovative signature for the development of cognitive dysfunction in hypertension. In particular, the effects of blood pressure variability and of different classes of antihypertensive drugs will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 40 and ≤ 70 years
* patients with moderate hypertension
* written informed consent

Exclusion Criteria:

* previous IMA, stroke or TIA
* arrhythmia or severe cardiac disease
* Diabetes or renal disease
* psychiatric disease
* neurological or neurodegenerative disease
* dementia
* assumption of drugs known to interfere with cognitive function
* inability to be subjected MRI analysis
* participation to other clinical trial, ongoing or terminated less than one month before enrolment in this study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients attending the Department of AngioCardioNeurology of the IRCCS Neuromed, accordingly to the following inclusion/exclusion criteria. Approximately 176 subjects of both genders will be included in the study.
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-12-08 (Estimated); Study Completion 2022-12-08 (Estimated)

PRIMARY OUTCOMES:
Measurement of percentage change in diffusion parameters of the white matter | At Enrollment; at 1 year Follow-up
  Fiber tracking by DTI MRI

SECONDARY OUTCOMES:
Detection of cognitive decline by decrease of MoCA score | At Enrollment; at 1 year Follow-up
  Cognitive tests
Characterization of cardiac hypertensive organ damage progression | At Enrollment; at 1 year Follow-up
  Echography
Characterization of renal hypertensive organ damage progression | At Enrollment; at 1 year Follow-up
  eGFR
Characterization of Blood Pressure Variability | At Enrollment; at 1 year Follow-up
  24h registration of systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No